CLINICAL TRIAL: NCT03276767
Title: An RCT Comparing Reminders Sendt by SMS or by E-mail in an Online Smoking Cessation Intervention
Brief Title: Comparing SMS and E-mail Reminders in an Online Smoking Cessation Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oslo (Other)
Collaborators: The Research Council of Norway (Other); Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Håvar Brendryen, Senior Research Scientist, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFR 228158/H10-C
Record Dates: First submitted 2017-09-07; First posted 2017-09-08 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Nicotine Dependence Tobacco Product
Keywords: online intervention; e-Health; reminder; SMS-textmessage; e-mail; mobile phone; cell phone
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants receive one out of two versions of a web-based smoking cessation program. The only difference between the two versions is the medium of the reminder: either SMS-textmessage or e-mail.
Masking Description: The recruitment procedure and the treatment is fully automated and delivered by web, e-mail and SMS-textmessages - i.e., the participant is not contacted by any care providers, investigators or assessors during recruitment or treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online intervention with SMS reminder (Experimental): Reminders will be sendt by SMS-TEXTMESSAGE if users of "Endre" does not log on to an assigned online session by noon on the second day.
  Interventions: Other: Endre
- Online intervention with e-mail reminder (Active Comparator): Reminder will be sendt by E-MAIL if users of "Endre" does not log on to an assigned online session by noon on the second day.
  Interventions: Other: Endre

INTERVENTIONS:
Other: Endre — The online intervention, "Endre", a digital smoking cessation counsellor that communicates with the user primarily through interactive web-sessions. Intervention content is tailored based on user input and individual usage pattern. Up to 14 unique sessions is assigned to the users during the study period, one each day. If a user does not start a session by noon on the second day a reminder will be sendt.

SUMMARY:
The primary purpose of the current study is to compare the effect of SMS-textmessage vs e-mail reminders on user engagement and proportion of reported quit attempts in an online smoking cessation intervention.

DETAILED DESCRIPTION:
Web- and mobile phone health behavior change interventions, including smoking cessation programs, offer great promise, but little is known about how such interventions should be designed to increase user engagement. The primary purpose of the current study is to compare the effect of SMS-textmessage vs e-mail reminders on user engagement and proportion of reported quit attempts in an online smoking cessation intervention.

The investigators propose a 2-arm RCT with 700 adult study participants that all receive a best practices web-based smoking cessation program designed for use on smart phones (web-app). The intervention includes a ten day preparation phase, in which participants continue smoking. On the eleventh day (and onward) the user will receive a session in which (s)he is asked whether (s)he has quit smoking or not. If not, the user will receive additional treatment sessions until (s)he reports having quit (or dropped out of the study). Each day (for up to 14 days) a new unique session is assigned to the user. However, if the user does not log on to the web-intervention and starts using the session by noon on the second day after assignment, the user will receive a reminder to do so. When a user is to be sent a reminder for the first time, (s)he will be randomized to either receive such reminders by SMS or by e-mail.

The primary outcome is reporting a quit attempt or not. Secondary outcomes include number web-sessions started and completed and time spent navigating sessions after the first reminder is received.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* current smoker
* determined to or considering to quit smoking
* provide valid e-mail address
* provide valid norwegian cell phone number
* complete a baseline questionnaire
* start using the intervention (pushing the next page button one time or more on the first session provided)
* has not logged on to any of the online session within noon on the second day after that particular session was made available

Exclusion Criteria:

* Not starting the first treatment session
* Taking every treatment session on time (no need for reminders, and thus not randomized)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2017-09-12 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Quit attempt | Within 6 weeks after starting the first session of the intervention
  User report a quit attempt

SECONDARY OUTCOMES:
Number of sessions completed | Within 6 weeks after starting the first session of the intervention
  Counted from after first reminder until reported quitting or study dropout (a unique session is made available each day)
Number of sessions started after first reminder | Within 6 weeks after starting the first session of the intervention
  Counted from after first reminder until reported quitting or study dropout (a unique session is made available each day)

CONTACTS AND LOCATIONS:
Overall Officials: Håvar Brendryen, PhD, Principal Investigator — University of Oslo
Locations (2):
- Department of Addictology, 1st Faculty of Medicine, Charles University, Prague, Czechia
- The Norwegian Centre for Addiction Research, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holter MT, Johansen A, Brendryen H. How a Fully Automated eHealth Program Simulates Three Therapeutic Processes: A Case Study. J Med Internet Res. 2016 Jun 28;18(6):e176. doi: 10.2196/jmir.5415. PMID 27354373
- [Derived] Kulhanek A, Lukavska K, Gabrhelik R, Novak D, Burda V, Prokop J, Holter MTS, Brendryen H. Comparing Reminders Sent via SMS Text Messaging and Email for Improving Adherence to an Electronic Health Program: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Mar 18;10(3):e31040. doi: 10.2196/31040. PMID 35302945
- See also: Web page of PI — https://www.sv.uio.no/psi/english/people/aca/haavabre/index.html